CLINICAL TRIAL: NCT05455554
Title: The Use of FlowMet-R Technology to Predict Wound Healing in Critical Limb Ischemia (CLI) Patients in a Wound Care Center Setting
Brief Title: The Use of FlowMet-R Technology to Predict Wound Healing in CLI Patients in a Wound Care Center Setting
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Stanford University (Other)
Collaborators: Medtronic Endovascular (Industry); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Venita Chandra, Clinical Associate Professor, Stanford University
Other Study IDs: 62133; 5R38HL143615-02 (NIH)
Record Dates: First submitted 2021-12-14; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- CLI (Critical Limb Ischemia): CLI cohort is a population of individuals with CLI, at least one active lower extremity wound and planned lower extremity revascularization. CLI cohort patients will receive Flowmet-D measurements in addition to standard of care therapy following intervention.
  Interventions: Diagnostic Test: Flowmet-D; Diagnostic Test: ABI
- HBO (Hyperbaric Oxygen): HBO cohort is a subset of the CLI cohort who will undergo hyperbaric oxygen therapy in the post-operative setting who will receive Flowmet-D measurements before and after their therapy.
  Interventions: Diagnostic Test: Flowmet-D; Diagnostic Test: ABI

INTERVENTIONS:
Diagnostic Test: Flowmet-D — Flowmet-D is a non-invasive device that measures blood flow.
Diagnostic Test: ABI — ABI is the ratio of the systolic blood pressure measured at the ankle to that measured at the brachial artery and is considered the gold standard for the diagnosis of peripheral artery disease.

SUMMARY:
Single-institution, prospective nonrandomized pilot study of critical limb ischemia patients with planned lower extremity revascularization will undergo Flowmet-D measurements in a wound care center setting to determine threshold values associated with wound healing and amputation. A subset of patients will undergo hyperbaric oxygen therapy and will have Flowmet-D measurements to determine those who respond best to therapy.

DETAILED DESCRIPTION:
A single-institution, prospective nonrandomized pilot study will be conducted at Stanford Hospital and the Stanford Advanced Wound Care Center (AWCC). Patients with CLTI by WIfI criteria (ABI or toe pressures) and a concomitant non-healing lower extremity wound will be recruited. Inclusion criteria will include CLTI, at least one active lower extremity wound and planned lower extremity revascularization. ABI/TBIs will be recorded preintervention, post intervention and at one and three month intervals. Intraprocedural characteristics including the number and location of vessels revascularized, patent runoff vessels pre and post procedure, pedal arch anatomy and presence of angiographic "blush" to wound will be documented.

Post-operatively, patients will be followed at the AWCC where they will receive standard of care wound management including offloading, regular debridement, infection and edema management. FlowMet-R perfusion values will be obtained prerevascularization, immediately post revascularization as well as weekly at each follow up AWCC visit for a total of up to 6 months or until wound healing.Wound size will be recorded.

Patients who undergo hyperbaric oxygen therapy (at the discretion of AWCC surgeon) will have perfusion values performed before and after hyperbaric oxygen therapy sessions 1, 2, 10, 20, 30 and 40. Hyperbaric oxygen therapy will be conducted 5 days a week for duration of 90 minutes. Patients who undergo other advanced wound care treatments such as stem cell therapies or skin substitutes will also received FlowMet-R prior to and after treatment. Primary outcomes will be wound healing defined as complete skin epithelialization, wound improvement rate, major and minor amputations as well as need for repeat revascularization.

ELIGIBILITY:
Inclusion Criteria:

CLI Cohort:

* CLI by WIfI criteria (ABI or toe pressures)
* Non-healing lower extremity wound
* Planned lower extremity revascularization
* Able to provide informed consent
* Able to comply with study procedures

HBO Cohort:

* All of the above
* Enrolled in HBO therapy post revascularization (at the discretion of the provider)

Exclusion Criteria:

* Under 30
* Wound not suitable for FlowMet-D probe attachment

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The CLI population is individuals with CLTI, at least one active lower extremity wound and planned lower extremity revascularization. The HBO cohort is a subset of the CLI population who will undergo HBO therapy post-revascularization.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-04-27 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Wound Healing | 6 months
  Wound Healing, defined as complete skin epithelialization, will be associated with Flowmet-D measurements.
Wound Improvement | 6 months
  Wound Improvement, defined as improvement in wound size, will be associated with Flowmet-D values.
Major Amputation | 6 months
  Major amputation, defined as amputation above the ankle joint, will be associated with Flowmet-D values.
Minor Amputation | 6 months
  Minor amputation, defined as amputation below the ankle joint, will be associated with Flowmet-D values.
Repeat Revascularization | 6 months
  Repeat Revascularization, defined as unplanned repeat lower extremity revascularization, will be monitored.

SECONDARY OUTCOMES:
Response to Hyperbaric Oxygen Therapy | 6 months
  Response to Hyperbaric Oxygen Therapy, will be defined as improved perfusion (improved Flowmet-D value) following therapy

CONTACTS AND LOCATIONS:
Overall Officials: Venita Chandra, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No